CLINICAL TRIAL: NCT04540666
Title: Sedation Sparing Effect of Virtual Reality in Third Molar Surgery
Brief Title: VR Sedation in Third Molar Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Chi-Wing, Clinical Doctor, Consultant of Department of Anaesthesiology, Queen Mary Hospital; Principal Investigator, Honorary Clinical Associate Professor, Department of Anaesthesiology, The University of Hong Kong, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UW20-453
Record Dates: First submitted 2020-08-27; First posted 2020-09-07 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia
Keywords: Anaesthesia for dental surgery; Sedation for dental surgery
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): VR program will be displayed throughout the surgery.
  Interventions: Drug: Propofol
- Non-VR group (Placebo Comparator): VR program will be turned off throughout the surgery.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Targeted Controlled Propofol Infusion will be set at 1 micro gram/ml.

SUMMARY:
Anaesthesia or sedation for dental surgery is Challenging. Over-sedation, leading to upper airway obstruction, desaturation and apnoea, is very common. On the other hand, it is also very common that inadequate sedative drugs were given, leading to under-sedation with unsatisfactory experience during operation. Therefore, it is good if some other methods are provided for sedation, avoiding side effects associated with sedative drugs.

DETAILED DESCRIPTION:
Immersive virtual reality (VR) is a form of distraction therapy and is believed to create an immersive experience that can restrict the mind from pain and anxiety and has been shown to be superior to simple distraction in reducing pain.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral impacted lower third molar that requires surgical removal
* Depth of impaction within 8mm as measured by Winter's line.
* Cantonese speaking

Exclusion Criteria:

* ASA > III
* BMI > 35
* Known Obstructive Sleep Apnoea
* Patients with known or potential difficult airway
* Chronic use of sedatives and opioid
* Alcohol or drug abuse
* Visual and hearing impairments
* Claustrophobia
* Cognitive impairment
* History of seizure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative propofol dose | From the start of anaesthesia to the end of anaesthesia, up to 2 hours after the start of surgery
  Amount of propofol required during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No